CLINICAL TRIAL: NCT01083706
Title: Treatment of Post-Transplant Relapse and Persistent Disease in Patients With MDS, CMML and AML With Azacitidine
Brief Title: Azacitidine in Treating Patients With Relapsed Myelodysplastic Syndrome, Chronic Myelomonocytic Leukemia, or Acute Myeloid Leukemia Who Have Undergone Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Bart Scott, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2240.00; NCI-2010-00281 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2240.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH); P01CA078902 (NIH)
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-04

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Childhood Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Myeloid Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes
MeSH Terms: conditions — Congenital Abnormalities; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemotherapy) (Experimental): Patients receive azacitidine SC or IV on days 1-7. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: azacitidine; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: azacitidine — Given SC or IV
  Other Names: 5-AC; 5-azacytidine; azacytidine; Vidaza
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well azacitidine works in treating patients with relapsed myelodysplastic syndrome (MDS), chronic myelomonocytic leukemia (CMML), or acute myeloid leukemia (AML) who have undergone stem cell transplant. Drugs used in chemotherapy, such as azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To improve overall survival in patients with post-transplant relapse of myeloid malignancies.

OUTLINE:

Patients receive azacitidine subcutaneously (SC) or intravenously (IV) on days 1-7. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* MDS, CMML or AML patients (as diagnosed by World Health Organization [WHO] criteria) with evidence of relapse or progression at >= day 28 and < day 100 post-transplant
* Recurrent or increased cytogenetic abnormalities by standard karyotype or fluorescence in situ hybridization (FISH) (the cytogenetic abnormalities must have been previously documented at some time point between diagnosis and date of stem cell transplant)
* Morphologic evidence of recurrence or increased abnormal myeloblasts in peripheral blood or marrow
* Flow Cytometric evidence of disease as determined by recurrent or increased abnormal myeloblasts in peripheral blood or marrow
* Extramedullary relapse (local radiotherapy will be allowed)
* MDS, CMML, or AML patients with persistent stable disease or persistent disease with regression at >= day 28 and < day 100 post-transplant; the inclusion of patients with persistent stable or persistent regressing disease in this protocol is not meant to advocate treatment; however, if the attending physician is inclined to offer treatment then these patients would be eligible for this study
* Persistence of cytogenetic abnormalities by standard karyotype or FISH
* Persistent morphologic evidence of abnormal myeloblasts (in patients with CMML the monoblastoid population is included) in peripheral blood or marrow
* Persistent flow cytometric evidence of abnormal myeloblasts (in patients with CMML the monoblastoid population is included) in peripheral blood or marrow
* Extramedullary persistence or regression

Exclusion Criteria:

* Refractory disease at time of stem cell transplant; patients who received chemotherapy prior to transplant with no evidence of response by International Working Group (IWG) criteria
* >= 10% bone marrow myeloblasts as measured by morphology
* Evidence of central nervous system (CNS) disease at time of relapse by morphology or flow (a diagnostic lumbar puncture [LP] is not required at time of relapse)
* Serum creatinine > 2 x ULN (upper limit of normal)
* Aspartate aminotransferase (AST)/ alanine aminotransferase (ALT) > 2x ULN
* Performance status > 2 (Eastern Cooperative Oncology Group [ECOG] Scale)
* Patients with severe disease other than MDS, CMML or AML which would be expected to prevent compliance with treatment
* Patients with severe infections (pneumonia, sepsis, etc) within the 2 weeks prior to the anticipated start of protocol treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-04; Primary Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Scott, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Chemotherapy)
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemotherapy)
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 52 [23 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 21

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Count of surviving participants at 6 months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy)
Number analyzed (Participants) | 39
Participants | 25

2. Secondary Outcome: Rate of Response by IWG Criteria
Description: Count of participants achieving a complete or partial remission at 6 months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy)
Number analyzed (Participants) | 39
Participants | 12

3. Secondary Outcome: Incidence of Grades II-IV Graft-versus-host Disease (GVHD)
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy)
Number analyzed (Participants) | 39
Participants | 25

ADVERSE EVENTS:
Arm/Group | Treatment (Chemotherapy)
Serious Adverse Events (participants affected / at risk) | 3/39
Other Adverse Events (participants affected / at risk) | 8/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy) (N=39)
Hospital Admission for Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hospital Admission for Cardioplumonary Arrest (Cardiac disorders) | 1 (1)
Hospital Admission for Cardioplumonary Arrest (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy) (N=39)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (11)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Infection- Rhizopus Pneumonia (Infections and infestations) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 2 (4)
Hypomagnesium (Metabolism and nutrition disorders) | 2 (3)
Elevated Billirubin (Metabolism and nutrition disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes